CLINICAL TRIAL: NCT05305365
Title: Phase IIa Study Assessing QBS72S For Treating Brain Metastases
Brief Title: Study Assessing QBS72S For Treating Brain Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Quadriga Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-63041; BRN0051 (Other: OnCore); NCI-2023-00648 (Other: CTRP)
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Brain Metastases; Breast Cancer; Lung Cancer; Leptomeningeal Disease; LMD
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms; Lung Neoplasms; Meningeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Patients with Breast Cancer Parenchymal brain metastasis (Cohort 1) (Experimental): All participants in Cohort 1 will receive QBS72S IV injections once monthly until disease progression.
  Interventions: Drug: QBS72S
- Patients with Breast Cancer Leptomeningeal Disease (Cohort 2) (Experimental): All participants in Cohort 2 will receive QBS72S IV injections once monthly until disease progression.
  Interventions: Drug: QBS72S
- Patients with any Primary Cancer Leptomeningeal Disease (Cohort 3) (Experimental): All participants in Cohort 3 will receive QBS72S IV injections once monthly until disease progression.
  Interventions: Drug: QBS72S

INTERVENTIONS:
Drug: QBS72S — QBS72S 18mg/m2 injection given intravenous once a month.
  Other Names: QBS10072S

SUMMARY:
This study is to evaluate the efficacy and safety of QBS72S in participants with advanced, relapsed, metastatic cancer with CNS involvement

DETAILED DESCRIPTION:
Primary Objective

1. Test of the preliminary efficacy of the intracranial anti tumor activity of QBS72S through overall response rate (ORR) in Cohort 1 (Stages 1+2).

Secondary Objectives

1. Test of the preliminary efficacy of the intracranial anti tumor activity of QBS72S through progression free survival (PFS) in Cohort 1 (Stages 1+2).
2. Test of the preliminary efficacy of the intracranial anti tumor activity of QBS72S through overall survival (OS) in Cohort 1 (Stages 1+2).
3. Test of the preliminary efficacy of the intracranial anti tumor activity of QBS72S through durations of response (DoR) in Cohort 1 (Stages 1+2).
4. Evaluate safety of QBS72S treatment in Cohort 1 (Stages 1+2), Cohort 2, and Cohort 3.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be 18 years or older
2. The participant must have a Karnofsky Performance Status (KPS) of 60 or above.
3. One of the following:

   1. Cohorts 1 and 2: The participant must have a histologically-confirmed breast cancer primary tumor, either confirmed via primary specimen or via metastasis site, having developed brain metastases (parenchymal or LMD) after a prior cytotoxic chemotherapy regimen.
   2. Cohort 3: The participant must have a histologically cancerous primary tumor, either confirmed via primary specimen or via metastasis site, having developed brain metastases (parenchymal or LMD) after a prior cytotoxic chemotherapy regimen. There is no restriction on prior cycles of systemic therapy for any primary cancer type. Breast cancer is not excluded from Cohort 3.
4. One of the following:

   1. Cohort 1: A participant with breast cancer brain parenchymal tumors must have at least one nonirradiated tumor ≥ 3 mm2 that can be seen on 2 or more separate acquired brain MRI sequences.
   2. Cohort 2: A participant with breast cancer primary and

   LMD must receive either:

   i. a brain MRI with contrast that supports the presence of LMD, or ii. a CSF cytology test that is either positive for or suspicious for malignancy. The presence of parenchymal brain metastases does not exclude these participants from Cohort 2.

   a. Cohort 3: A participant with LMD from any primary cancer site must receive either: i. a brain MRI with contrast that supports the presence of LMD, or ii. a CSF cytology test that is either positive for or suspicious for malignancy. The presence of parenchymal brain metastases does not exclude these participants from Cohort 3.
5. For corticosteroids and anticonvulsants, the participant must either: c. not be taking any, or d. be taking stable or decreasing doses for ≥5 days prior to obtaining the screening Gd-MRI of the brain. The maximum allowable dose of corticosteroids is 8mg of dexamethasone per day, or the equivalent of another medication as assessed by a Neuro-Oncologist. Escalation of corticosteroids is not allowed ≤14 days prior to C1D1.
6. The participant must have completed washout from prior therapy before C1D1, as applicable: e. ≥7 days for Ommaya placement (Cohorts 2+3) f. ≥14 days for small molecules and non-cytotoxic systemic drugs e.g., PARP inhibitors g. ≥21 days for checkpoint inhibitors and monoclonal antibodies, e.g., atezolizumab, pembrolizumab, and bevacizumab, and cytotoxic chemotherapy h. ≥28 days for investigational drugs, radiotherapy, and major surgery. Minor procedures such as tumor biopsy are allowed with written approval from the PI i. ≥1 dosing cycle for other interventions All significant toxicities from previous anticancer therapy must have stabilized to a new baseline or have resolved. Participation in long term follow up in another clinical trial is allowed if no procedures will be performed which may interfere with the interpretation of study results.
7. The participant must have adequate bone marrow function, including: j. ANC ≥ 1,500/mm3 or ≥ 1.5 x 109/L k. Platelets ≥ 100,000/ mm3 or ≥ 100 x 109/L l. Hemoglobin ≥ 9 g/dL
8. The participant must have adequate renal function, including serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 50 mL/min. In equivocal cases, a 24-hour urine collection test can be used to estimate the creatinine clearance more accurately.
9. The participant must have adequate liver function, including: m. Total serum bilirubin ≤ 1.5 x ULN unless the participant has documented Gilbert syndrome who must have a total bilirubin < 3.0 mg/dl n. Aspartate and Alanine aminotransferase (AST and ALT) ≤ 2.5 x ULN; ≤ 5.0 x ULN if there is liver involvement by the tumor
10. Any participant physiologically capable of becoming pregnant or getting a partner pregnant must agree to use highly effective contraception during study treatment and for 7 months after study discontinuation.
11. Participants or their designated advocates must be willing to and capable of providing informed consent and willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures

Exclusion Criteria

1. Participants with any other current, active malignancy unrelated to their primary cancer diagnosis, except for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ.
2. Participants with intolerance to or who have had a severe (Grade 3) allergic or anaphylactic reaction to any of the substances included in the investigational product: sulfobutylether-β-cyclodextrin, melphalan, bendamustine, chlorambucil or any nitrogen mustard chemotherapeutics.
3. Participants who currently use or have an anticipated need for a contraindicated medication including live vaccines, natalizumab, nivolumab, ocrelizumab, palifermin, pimecrolimus, tacrolimus, tofacitinib, and EIAEDs, including phenytoin, phenobarbital, carbamazepine, fosphenytoin, primidone, and oxcarbazepine. The washout period for any live vaccine is 30 days prior to enrollment. There is no restriction for seasonal flu vaccines that do not contain live virus, nor any approved COVID vaccine.
4. Participants who are pregnant or breastfeeding.
5. Participants who have active medical or psychiatric conditions which, in the opinion of the Principal Investigator or a Sub-Investigator, would compromise or interfere with their ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response against Intracranial Tumor Lesions, Cohort 1 (Stages 1+2) | 6 months
  The overall response against the target intracranial tumor lesions in Cohort 1 (Stages 1+2) participants was assessed by according to the modified Response Assessment in Neuro-oncology for Brain Metastases (mRANO-BM)
RECIST 1.1 response criteria | 6 months from the start of treatment
  Clinical response means either a complete response (CR) or a partial response (PR). CR is defined as disappearance of tumor lesions, and PR is defined as ≥ 30% reduction in diameter of tumor lesions.

SECONDARY OUTCOMES:
Progression-free Survival (PFS), Cohort 1 (Stages 1+2) | 2 months
  Progression-free Survival (PFS) means to remain alive without tumor progression, assessed as a ≥ 25% increase in tumor diameter
Overall Survival (OS), Cohort 1 (Stages 1+2) | 2 months
  Overall survival (OS) refers to remaining alive at the time of the assessment.
Duration of Response (DoR), Cohort 1 (Stages 1+2) | 6 months
  Duration of Response (DoR) refers to length of time that a clinical response is maintained in Cohort 1 (Stages 1+2) participants.
Related Adverse Events (AEs) | 30 days following the last administration of study drug
  Toxicity refers to drug-related adverse events (AEs). The outcome is reported as the number of related AEs that were serious or non-serious, and by severity (mild, moderate, severe, life-threatening, or fatal), numbers without dispersion

CONTACTS AND LOCATIONS:
Overall Officials: Melanie H Gephart, MD, MAS, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Institute, Palo Alto, California, United States

REFERENCES:
- [Derived] Taiwo R, Harary PM, Trinh TTH, Granucci M, Bertrand S, Carlson-Clarke B, Chernikova SB, Therkelsen K, Arora M, Melisko ME, Iv M, Vogel H, Han S, Xie C, Brain S, Lee V, Bharani KL, Nagpal S, Hayden Gephart M. Adaptive cohort design and LAT1 expression scale: study protocol for a Phase 2a trial of QBS72S in breast cancer brain metastases. BMC Cancer. 2025 Aug 15;25(1):1316. doi: 10.1186/s12885-025-14282-x. PMID 40813655